CLINICAL TRIAL: NCT06424353
Title: Postoperative Pain After Pulpectomy of Primary Molars Using Two Different Root Canal Obturation Techniques: A Randomized Clinical Trial
Brief Title: Postoperative Pain After Pulpectomy of Primary Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Abdel Hafeez, postgraduate student at faculty of dentistry, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 87-577
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lentilospiral group (Experimental): Obturation of primary molars with calcium hydroxide, eugenol and iodoform paste using paste carrier files(lentiospiral files)
  Interventions: Procedure: Endoflas pulpectomy
- pressure seringe group (Active Comparator): Obturation of primary molars with calcium hydroxide, eugenol and iodoform paste using pressure seringe
  Interventions: Procedure: Endoflas pulpectomy

INTERVENTIONS:
Procedure: Endoflas pulpectomy — obturation of root canals of primary molars with Endoflas using pressure seringe and lentilospiral files

SUMMARY:
Testing postopertive pain after pulpectomy of primary molars with endoflas using modified Wong-Baker scale of pain.

DETAILED DESCRIPTION:
Testing postopertive pain after pulpectomy of primary molars with endoflas using lentilospiral files and pressure seringe by using modified Wong-Baker scale of pain.

ELIGIBILITY:
Inclusion Criteria:

* The current study will include children who meet the following clinical and radiographic criteria:

3.1a.Clinical:

1. 5-7-year old children categorized as class I or II according to American Society of Anaesthesiologists (ASA) scale.
2. Children rated as no.3 or 4 in Frankel behavior rating scale (FBRS).
3. Presence of at least one primary molar with deep carious lesion.
4. Asymptomatic necrotic molars confirmed by the absence of bleeding on opening of the pulp chamber.

3.1b. Radiographic:

1. Extensive caries approaching to the pulp.
2. Presence of at least two-thirds of root length.

Exclusion Criteria:

* A child's tooth with any of the following criteria:

3.2a. Clinical findings:

1. History of spontaneous unprovoked toothache.
2. Extensive crown destruction that preclude coronal restoration.
3. Presence of adjacent or opposing tooth with deep carious lesion "in the same side".
4. History of administering analgesics 12 hours before tooth obturation.

3.2b. Radiographic findings:

1. Presence of a large furcation or periapical radiolucency approximating the succedaneous tooth.
2. Presence of pathological internal/external root resorption.
3. Absence of underlying permanent successor.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | after one day and after one week
  Measuring post operative pain after pulpectomy with two different obturation techniques using (Modified Wong-backer scale of pain )which have four scales from( 0 to 3) which 0 is the better outcome( no pain) and 3 is the worst (severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: osama s gad elhak, phD, Study Director — Pediatric Dentistry Department, Faculty of Dentistry, Minia University
Locations (1):
- Shimaa Mohamed Abd Elhafeez, Minya, Egypt